CLINICAL TRIAL: NCT03128411
Title: A PHASE 2, OPEN-LABEL, SINGLE-ARM STUDY TO EVALUATE EFFICACY AND SAFETY OF BOSUTINIB MONOTHERAPY IN JAPANESE ADULT PATIENTS WITH NEWLY DIAGNOSED CHRONIC PHASE CHRONIC MYELOGENOUS LEUKEMIA
Brief Title: Study of Bosutinib in Japanese Adult Patients With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1871048
Record Dates: First submitted 2017-03-28; First posted 2017-04-25 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: Leukemia, Chronic Myelogenous
Keywords: Leukemia, Chronic Myelogenous
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bosutinib (Experimental): Bosutinib monotherapy; All patients will receive bosutinib at a starting dose of 400 mg QD. The dose of bosutinib may be escalated (up to a maximum of 600 mg QD) for unsatisfactory response or reduced for toxicity.
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — All patients will receive bosutinib at a starting dose of 400 mg QD.

SUMMARY:
Phase 2, single-arm, open-label trial. Patients will receive bosutinib for the duration of the study.

DETAILED DESCRIPTION:
The study will be open for enrollment until the planned number of approximately 60 Philadelphia Chromosome Positive (Ph+) patients have been registered. All patients will be treated and/or followed for up to approximately 3 years (144 weeks) after registration of the last patient or until study termination. Patients who discontinue study therapy early due to disease progression or intolerance to study medication will continue to be followed yearly for survival for up to approximately 3 years (144 weeks) after registration of the last patient or until study termination.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP CML of ≤6 months (from initial diagnosis); Diagnosis of CP CML with molecular confirmation by detection of BCR-ABL rearrangement at screening (cytogenetic assessment for Ph is not required for enrollment; however, patients with known Ph- CML prior to registration are not eligible for this study)
* Age ≥20 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Adequate Liver and Renal Function

Exclusion Criteria:

* Any prior medical treatment for CML, including TKIs, with the exception of hydroxyurea treatment, which is permitted for up to 6 months prior to registration
* Any past or current CNS involvement, including leptomeningeal leukemia
* Extramedullary disease only
* Major surgery or radiotherapy within 14 days prior to registration
* History of clinically significant or uncontrolled cardiac disease
* Patients with active, uncontrolled bacterial, fungal, or viral infection
* Recent or ongoing clinically significant GI disorder
* History of another malignancy within 5 years prior to registration
* Uncontrolled hypomagnesemia or uncorrected hypokalemia due to potential effects on the QT interval
* Known prior or suspected severe hypersensitivity to study drugs or any component in their formulations
* Participation in other studies involving investigational drug(s) within 30 days or 5 half-lives of investigational product, whichever is longer, prior to registration and/or during study participation
* Other severe acute or chronic medical or psychiatric condition, including recent or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or interfere with the interpretation of study results
* Investigational site staff members directly involved in the conduct of the study and their family members, or Pfizer employees, including their family members, directly involved in the conduct of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- Japan (21):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - Japanese Red Cross Narita Hospital, Narita, Chiba
  - Ehime University Hospital, Toon-shi, Ehime
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Osaka City University Hospital, Osaka, Osaka
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyo-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - Chiba University Hospital, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Saga University Hospital, Saga
  - Nippon Medical School Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Garrett M, Knight B, Cortes JE, Deininger MW. Population modeling of bosutinib exposure-response in patients with newly diagnosed chronic phase chronic myeloid leukemia. Cancer Med. 2023 Sep;12(17):17981-17992. doi: 10.1002/cam4.6439. Epub 2023 Aug 8. PMID 37553873
- [Derived] Ono T, Hino M, Matsumura I, Fujisawa S, Ishizawa K, Sakaida E, Sekiguchi N, Ono C, Aizawa M, Tanetsugu Y, Koide Y, Takahashi N. Bosutinib in Japanese patients with newly diagnosed chronic-phase chronic myeloid leukemia: final 3-year follow-up results of a phase 2 study. Int J Hematol. 2022 Dec;116(6):871-882. doi: 10.1007/s12185-022-03435-4. Epub 2022 Aug 13. PMID 35963986
- [Derived] Takahashi N, Cortes JE, Sakaida E, Ishizawa K, Ono T, Doki N, Matsumura I, Garcia-Gutierrez V, Rosti G, Ono C, Ohkura M, Tanetsugu Y, Viqueira A, Brummendorf TH. Safety profile of bosutinib in Japanese versus non-Japanese patients with chronic myeloid leukemia: a pooled analysis. Int J Hematol. 2022 Jun;115(6):838-851. doi: 10.1007/s12185-022-03314-y. Epub 2022 Mar 2. PMID 35235189
- [Derived] Hino M, Matsumura I, Fujisawa S, Ishizawa K, Ono T, Sakaida E, Sekiguchi N, Tanetsugu Y, Fukuhara K, Ohkura M, Koide Y, Takahashi N. Phase 2 study of bosutinib in Japanese patients with newly diagnosed chronic phase chronic myeloid leukemia. Int J Hematol. 2020 Jul;112(1):24-32. doi: 10.1007/s12185-020-02878-x. Epub 2020 Apr 11. PMID 32279228
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1871048

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosutinib: Participants with newly diagnosed CP CML received bosutinib treatment, orally at a dose of 400 mg QD. In treatment phase, participants received bosutinib once daily for up to 12 months, which was extended further to at least additional 24 months (total of at least 36 months) or until end of the study, treatment failure, unacceptable toxicity, death, or withdrawal of consent, whichever occurred first. If participants discontinued the treatment phase only then they entered the long-term follow-up phase up to approximately 3 years after registration of the last participant, or until study termination, whichever comes first.
Period: Treatment Phase
Arm/Group | Bosutinib
Started | 60
Received Treatment | 60
Completed | 36
Not Completed | 24
Not completed — Adverse Event | 21
Not completed — Physician Decision | 1
Not completed — Other | 2
Period: Long Term Follow-up Phase
Arm/Group | Bosutinib
Started | 24 (Participants who discontinued treatment phase, entered in long term follow up phase.)
Completed | 22
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: As-treated population included all enrolled participants who received at least 1 dose of study treatment.
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (16.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 60
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Molecular Response (MMR) at Month 12
Description: A MMR is defined as less than or equal to (<=) 0.1 percent (%) BCR-ABL transcripts on the international scale (IS), corresponding to a >=3-log reduction from standardized baseline with at least 3000 ABL assessed by the central laboratory. The MMR value counted only if the response was demonstrated at the 12-month visit; any MMR gained and lost, or never achieved at or before the 12-month visit was considered as non-responder.
Time Frame: Month 12
Population: The modified as-treated population included all enrolled participants with Philadelphia chromosome positive CP CML harboring b2a2 and/or b3a2 transcripts who received at least 1 dose of study treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 55.0 [44.4 to 65.6]
Statistical Analysis 1: Comparison: Bosutinib; With a sample size of 60 participants, study was powered at >82% to test null hypothesis: true MMR rate at 12 months (48 weeks) is 25% versus alternative hypothesis: true MMR rate is 40% with one-sided alpha of 5%; Test type: Superiority; p < 0.0001, z-test, 1-sided

2. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) by Month 12
Description: A MMR is defined as less than or equal to (<=) 0.1 percent (%) BCR-ABL transcripts on the international scale (IS), corresponding to a >=3-log reduction from standardized baseline with at least 3000 ABL assessed by the central laboratory. The MMR value counted only if the response was demonstrated at or before the 12-month visit.
Time Frame: Up to Month 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 61.7 [51.3 to 72.0]

3. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) by Month 18
Description: A MMR is defined as less than or equal to (<=) 0.1 percent (%) BCR-ABL transcripts on the international scale (IS), corresponding to a >=3-log reduction from standardized baseline with at least 3000 ABL assessed by the central laboratory. The MMR value counted only if the response was demonstrated at or before the 18-month visit.
Time Frame: Up to Month 18
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 66.7 [56.7 to 76.7]

4. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR) by Month 12
Description: CCyR is based on the prevalence of Philadelphia chromosome positive metaphases among cells in metaphase on a bone marrow sample. CCyR was defined as absence of detectable Philadelphia chromosome positive cells. CCyR was achieved when there were "0" Philadelphia chromosome positive metaphases among at least 20 metaphases from a bone marrow sample or when MMR was achieved if no bone marrow analysis was performed. The CCyR value was counted only if the response was demonstrated at or before the 12-month visit.
Time Frame: Up to Month 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 80.0 [71.5 to 88.5]

5. Secondary Outcome: Probability of Maintaining Major Molecular Response (MMR) at Month 36
Description: Duration of MMR: time from first date of MMR until first date of confirmed loss of MMR, treatment discontinuation due to progressive disease (PD), or death due to PD within 28 days after last dose or censoring. PD: progression to Accelerated phase (AP) or to Blast Phase (BP). AP: 15-29% blasts in blood or marrow, or>30% blasts plus promyelocytes in blood or marrow with blasts <30%; ≥20% basophils in blood. BP: ≥30% Blasts in blood or bone marrow, extramedullary blast proliferation, other than in spleen. Kaplan-Meier analysis was used.
Time Frame: At Month 36
Population: The modified as-treated population included all enrolled participants with Philadelphia chromosome positive CP CML harboring b2a2 and/or b3a2 transcripts who received at least 1 dose of study treatment. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure and who had MMR.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 42
Percentage of participants | 100.0 [100.0 to 100.0]

6. Secondary Outcome: Probability of Maintaining Complete Cytogenetic Response (CCyR) at Month 36
Description: Duration of CCyR, from first date of CCyR to confirmed loss of CCyR, treatment discontinuation due to PD, death due to PD within 28 days after last dose or censoring. Confirmed loss: at least 1 Ph+ metaphase confirmed by a second determination >=4 weeks later or unconfirmed loss followed by treatment discontinuation due to suboptimal response. PD: progression to AP or to BP. Kaplan-Meier analysis was used.
Time Frame: At Month 36
Population: The modified as-treated population included all enrolled participants with Philadelphia chromosome positive CP CML harboring b2a2 and/or b3a2 transcripts who received at least 1 dose of study treatment. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure and who had CCyR.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 48
Percentage of participants | 100.0 [100.0 to 100.0]

7. Secondary Outcome: Cumulative Incidence of Event Free Survival (EFS) at Month 36
Description: EFS: time from 1st dose until 1st occurrence of 1 of the following events or censoring: 1)death from any cause 2)transformation to AP or BP 3)loss of complete hematologic response (CHR) 4)loss of CCyR 5)participants not achieving CHR: doubling of WBCs >= 1 month apart with 2nd value >20*10^9/L and maintained in subsequent assessments for >=2 weeks. Loss of CHR: appearance of any of the following confirmed by 2nd determination>=4 weeks later (unless associated with CML-related treatment discontinuation): WBC count: >20.0*10^9/L, platelet count: >=600*10^9/L, appearance of palpable spleen/other extra medullary involvement, appearance of 5% myelocytes or blasts or promyelocytes in peripheral blood. Loss of CCyR:>= one Ph+ metaphase confirmed by 2nd determination >=4 weeks later(unless associated with CML-related treatment discontinuation). Cumulative incidence: % of participants with event at month 36 adjusted for competing risk of treatment discontinuation without event.
Time Frame: Up to Month 36
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 1.7 [0.2 to 6.4]

8. Secondary Outcome: Probability of Overall Survival (OS) at Month 36
Description: Overall survival was defined as the time from first dose of study drug to death due to any cause or censoring. Kaplan-Meier analysis was used for determination of probability of overall survival.
Time Frame: Up to Month 36
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 96.7 [89.7 to 98.9]

9. Secondary Outcome: Trough Plasma Concentrations of Bosutinib
Time Frame: Pre-dose on Day 1, Day 28, Day 56, Day 84
Population: The PK population will be defined as any patient in the safety population of patients who had at least 1 concentration of bosutinib on-treatment.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Nanogram per milliliter (ng/mL)
  Day 1 | 0.000 (0.000)
  Day 28: number analyzed (Participants) | 34
  Day 28 | 83.564 (64.1056)
  Day 56: number analyzed (Participants) | 41
  Day 56 | 85.963 (46.4095)
  Day 84: number analyzed (Participants) | 44
  Day 84 | 79.659 (41.5369)

10. Secondary Outcome: Summary and Analysis of Trough Bosutinib Plasma Concentration by Major Molecular Response (MMR) Response
Description: Trough bosutinib plasma concentration is reported classified on basis of participants with MMR response as "Yes" and "No" at specified time points. A MMR is defined as less than or equal to (<=) 0.1 percent (%) BCR-ABL transcripts on the international scale (IS), corresponding to a >=3-log reduction from standardized baseline with at least 3000 ABL assessed by the central laboratory.
Time Frame: Pre-dose on Day 28, Day 56 and Day 84
Population: PK population included of all enrolled participants, who received at least 1 dose of study treatment and had at least 1 concentration of bosutinib on-treatment. For Day 28, 56, 84: total number of participants analyzed for each time point were sum of "number analyzed" against Yes and No categories respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Yes: Day 28: number analyzed (Participants) | 23
  Yes: Day 28 | 94.943 (71.9332)
  No: Day 28: number analyzed (Participants) | 11
  No: Day 28 | 59.770 (35.4568)
  Yes: Day 56: number analyzed (Participants) | 26
  Yes: Day 56 | 88.196 (48.9671)
  No: Day 56: number analyzed (Participants) | 15
  No: Day 56 | 82.092 (42.9741)
  Yes: Day 84: number analyzed (Participants) | 31
  Yes: Day 84 | 81.339 (41.5443)
  No: Day 84: number analyzed (Participants) | 13
  No: Day 84 | 75.654 (42.9290)

11. Secondary Outcome: Summary and Analysis of Trough Bosutinib Plasma Concentration by CCyR Response
Description: Trough bosutinib plasma concentration is reported classified on basis of participants with CCyR Response as "Yes" and "No" at specified time points. CCyR is based on the prevalence of Philadelphia chromosome positive metaphases among cells in metaphase on a bone marrow sample. CCyR was defined as absence of detectable Philadelphia chromosome positive cells. CCyR was achieved when there were "0" Philadelphia chromosome positive metaphases among at least 20 metaphases from a bone marrow sample or when MMR was achieved if no bone marrow analysis was performed.
Time Frame: Pre-dose on Day 28, Day 56 and Day 84
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Yes: Day 28: number analyzed (Participants) | 32
  Yes: Day 28 | 87.006 (64.1820)
  No: Day 28: number analyzed (Participants) | 2
  No: Day 28 | 28.490 (38.3393)
  Yes: Day 56: number analyzed (Participants) | 36
  Yes: Day 56 | 90.550 (45.4543)
  No: Day 56: number analyzed (Participants) | 5
  No: Day 56 | 52.936 (43.6721)
  Yes: Day 84: number analyzed (Participants) | 41
  Yes: Day 84 | 79.429 (40.1538)
  No: Day 84: number analyzed (Participants) | 3
  No: Day 84 | 82.800 (69.5117)

12. Secondary Outcome: Summary of Trough Bosutinib Plasma Concentration by Total Bilirubin
Description: Trough bosutinib plasma concentration is reported classified on basis of total bilirubin level range at baseline. Level range 1: <=7.7 micromole per liter (micromol/L), level rage 2: >7.7 and <= 10.3 micromol/L, level range 3: >10.3 and <=12.85 micromol/L and level range 4: >12.85 micromol/L.
Time Frame: Pre-dose on Day 28, Day 56 and Day 84
Population: PK population included of all enrolled participants, who received at least 1 dose of study treatment and had at least 1 concentration of bosutinib on-treatment. For Day 28, 56, 84: total number of participants analyzed for each time point were sum of "number analyzed" against each categories/levels respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Day 28: (<=7.7 micromol/L): number analyzed (Participants) | 6
  Day 28: (<=7.7 micromol/L) | 61.833 (18.0632)
  Day 28: (>7.7 and <=10.3 micromol/L): number analyzed (Participants) | 12
  Day 28: (>7.7 and <=10.3 micromol/L) | 96.867 (87.7756)
  Day 28: (>10.3 and <=12.85 micromol/L): number analyzed (Participants) | 6
  Day 28: (>10.3 and <=12.85 micromol/L) | 76.963 (59.0962)
  Day 28: (>12.85 micromol/L): number analyzed (Participants) | 10
  Day 28: (>12.85 micromol/L) | 84.599 (54.3057)
  Day 56: (<=7.7 micromol/L): number analyzed (Participants) | 9
  Day 56: (<=7.7 micromol/L) | 60.044 (22.6753)
  Day 56: (>7.7 and <=10.3 micromol/L): number analyzed (Participants) | 13
  Day 56: (>7.7 and <=10.3 micromol/L) | 81.246 (44.3985)
  Day 56: (>10.3 and <=12.85 micromol/L): number analyzed (Participants) | 7
  Day 56: (>10.3 and <=12.85 micromol/L) | 91.940 (49.9495)
  Day 56: (>12.85 micromol/L): number analyzed (Participants) | 12
  Day 56: (>12.85 micromol/L) | 107.025 (53.5192)
  Day 84: (<=7.7 micromol/L): number analyzed (Participants) | 8
  Day 84: (<=7.7 micromol/L) | 50.775 (19.4910)
  Day 84: (>7.7 and <=10.3 micromol/L): number analyzed (Participants) | 18
  Day 84: (>7.7 and <=10.3 micromol/L) | 75.478 (34.0806)
  Day 84: (>10.3 and <=12.85 micromol/L): number analyzed (Participants) | 6
  Day 84: (>10.3 and <=12.85 micromol/L) | 98.133 (56.5691)
  Day 84: (>12.85 micromol/L): number analyzed (Participants) | 12
  Day 84: (>12.85 micromol/L) | 95.950 (46.2820)

13. Secondary Outcome: Summary of Trough Bosutinib Plasma Concentration by Creatinine Clearance
Description: Trough bosutinib plasma concentration is reported classified on basis of different ranges of creatinine clearance at baseline. Level range 1: <=71.479 milliliter per minute (mL/min), level rage 2: >71.479 and <=100.936 mL/min, level range 3: >100.936 and <=129.355 mL/min) and level range 4: >129.355 mL/min.
Time Frame: Pre-dose on Day 28, Day 56 and Day 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Day 28: (<=71.479 mL/min): number analyzed (Participants) | 7
  Day 28: (<=71.479 mL/min) | 75.039 (63.7599)
  Day 28: (>71.479 and <=10 0.936 mL/min): number analyzed (Participants) | 7
  Day 28: (>71.479 and <=10 0.936 mL/min) | 84.114 (49.0390)
  Day 28: (>100.936 and <=1 29.355 mL/min): number analyzed (Participants) | 10
  Day 28: (>100.936 and <=1 29.355 mL/min) | 100.100 (97.8388)
  Day 28: (>129.355 mL/min): number analyzed (Participants) | 10
  Day 28: (>129.355 mL/min) | 72.610 (26.2392)
  Day 56:(<=71.479 mL/min): number analyzed (Participants) | 5
  Day 56:(<=71.479 mL/min) | 93.056 (56.2220)
  Day 56:(>71.479 and <=10 0.936 mL/min): number analyzed (Participants) | 11
  Day 56:(>71.479 and <=10 0.936 mL/min) | 92.764 (47.9905)
  Day 56: (>100.936 and <=1 29.355 mL/min): number analyzed (Participants) | 10
  Day 56: (>100.936 and <=1 29.355 mL/min) | 95.580 (58.4145)
  Day 56: (>129.355 mL/min): number analyzed (Participants) | 15
  Day 56: (>129.355 mL/min) | 72.200 (32.9961)
  Day 84: (<=71.479 mL/min): number analyzed (Participants) | 10
  Day 84: (<=71.479 mL/min) | 92.540 (49.2182)
  Day 84:(>71.479 and <=10 0.936 mL/min): number analyzed (Participants) | 10
  Day 84:(>71.479 and <=10 0.936 mL/min) | 90.590 (45.9533)
  Day 84:(>100.936 and <=1 29.355 mL/min): number analyzed (Participants) | 11
  Day 84:(>100.936 and <=1 29.355 mL/min) | 69.100 (41.0767)
  Day 84: (>129.355 mL/min): number analyzed (Participants) | 13
  Day 84: (>129.355 mL/min) | 70.277 (30.6643)

14. Secondary Outcome: Summary of Trough Bosutinib Plasma Concentration by Aspartate Aminotransferase
Description: Trough bosutinib plasma concentration is reported classified on basis of different ranges of aspartate aminotransferase at baseline. Level range 1: <=22 units per liter (U/L), level rage 2: >22 and <=26 U/L, level range 3: >26 and <=33 U/L and level range 4: >33 U/L.
Time Frame: Pre-dose on Day 28, Day 56 and Day 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Day 28: (<=22 U/L): number analyzed (Participants) | 7
  Day 28: (<=22 U/L) | 65.771 (26.3239)
  Day 28: (>22 and <=26 U/L): number analyzed (Participants) | 6
  Day 28: (>22 and <=26 U/L) | 140.617 (120.1651)
  Day 28: (>26 and <=33 U/L): number analyzed (Participants) | 12
  Day 28: (>26 and <=33 U/L) | 66.056 (37.4551)
  Day 28: (>33 U/L): number analyzed (Participants) | 9
  Day 28: (>33 U/L) | 82.711 (47.9527)
  Day 56: (<=22 U/L): number analyzed (Participants) | 12
  Day 56: (<=22 U/L) | 82.117 (51.0937)
  Day 56: (>22 and <=26 U/L): number analyzed (Participants) | 8
  Day 56: (>22 and <=26 U/L) | 76.050 (43.6907)
  Day 56: (>26 and <=33 U/L): number analyzed (Participants) | 12
  Day 56: (>26 and <=33 U/L) | 93.607 (44.5087)
  Day 56: (>33 U/L): number analyzed (Participants) | 9
  Day 56: (>33 U/L) | 89.711 (50.6123)
  Day 84: (<=22 U/L): number analyzed (Participants) | 10
  Day 84: (<=22 U/L) | 54.550 (23.4932)
  Day 84: (>22 and <=26 U/L): number analyzed (Participants) | 8
  Day 84: (>22 and <=26 U/L) | 81.325 (55.3891)
  Day 84: (>26 and <=33 U/L): number analyzed (Participants) | 14
  Day 84: (>26 and <=33 U/L) | 85.886 (39.3348)
  Day 84: (>33 U/L): number analyzed (Participants) | 12
  Day 84: (>33 U/L) | 92.208 (41.4203)

15. Secondary Outcome: Summary of Trough Bosutinib Plasma Concentration by Alanine Aminotransferase
Description: Trough bosutinib plasma concentration is reported classified on basis of different ranges of alanine aminotransferase at baseline. Level range 1: <=17.5 U/L, level rage 2: >17.5 and <=25 U/L, level range 3: >25 and <=32 U/L and level range 4: >32 U/L.
Time Frame: Pre-dose on Day 28, Day 56 and Day 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Day 28: (<=17.5 U/L): number analyzed (Participants) | 7
  Day 28: (<=17.5 U/L) | 49.111 (24.6077)
  Day 28: (>17.5 and <=25 U/L): number analyzed (Participants) | 6
  Day 28: (>17.5 and <=25 U/L) | 98.882 (131.3382)
  Day 28: (>25 and <=32 U/L): number analyzed (Participants) | 12
  Day 28: (>25 and <=32 U/L) | 94.175 (44.7227)
  Day 28: (>32 U/L): number analyzed (Participants) | 9
  Day 28: (>32 U/L) | 86.000 (39.7021)
  Day 56: (<=17.5 U/L): number analyzed (Participants) | 10
  Day 56: (<=17.5 U/L) | 66.878 (33.4154)
  Day 56: (>17.5 and <=25 U/L): number analyzed (Participants) | 6
  Day 56: (>17.5 and <=25 U/L) | 82.317 (69.6971)
  Day 56: (>25 and <= 32 U/L): number analyzed (Participants) | 12
  Day 56: (>25 and <= 32 U/L) | 104.350 (47.3634)
  Day 56: (>32 U/L): number analyzed (Participants) | 13
  Day 56: (>32 U/L) | 85.354 (40.1619)
  Day 84: (<=17.5 U/L): number analyzed (Participants) | 9
  Day 84: (<=17.5 U/L) | 65.011 (43.4694)
  Day 84: (>17.5 and <=25 U/L): number analyzed (Participants) | 9
  Day 84: (>17.5 and <=25 U/L) | 73.511 (43.4070)
  Day 84: (>25 and <=32 U/L): number analyzed (Participants) | 13
  Day 84: (>25 and <=32 U/L) | 92.254 (49.1564)
  Day 84: (>32 U/L): number analyzed (Participants) | 13
  Day 84: (>32 U/L) | 81.462 (29.7583)

16. Secondary Outcome: Summary and Analysis of Trough Bosutinib Plasma Levels by Presence/Absence Grade 1: Diarrhea
Description: Trough bosutinib plasma concentration is reported classified on basis of presence/ or absence of grade 1 diarrhea as "Yes" and "No" at specified time points. As per national cancer institute common terminology criteria (NCI-CTCAE) version 4.03, Grade 1: increase of <4 stools per day over baseline.
Time Frame: Pre-dose on Day 28, Day 56 and Day 84 for trough bosutinib plasma concentration up to 12 March 2019; maximum of 22 months, approximately, for the adverse event of interest
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Yes: Day 28: number analyzed (Participants) | 28
  Yes: Day 28 | 85.585 (69.4219)
  No: Day 28: number analyzed (Participants) | 6
  No: Day 28 | 74.133 (31.1208)
  Yes: Day 56: number analyzed (Participants) | 36
  Yes: Day 56 | 86.086 (46.9140)
  No: Day 56: number analyzed (Participants) | 5
  No: Day 56 | 85.080 (47.7414)
  Yes: Day 84: number analyzed (Participants) | 37
  Yes: Day 84 | 85.219 (41.7195)
  No: Day 84: number analyzed (Participants) | 7
  No: Day 84 | 50.271 (26.8976)

17. Secondary Outcome: Summary and Analysis of Trough Bosutinib Plasma Levels by Presence/Absence Grade 1: Nausea
Description: Trough bosutinib plasma concentration is reported classified on basis of presence/ or absence of grade 1 Nausea as "Yes" and "No" at specified time points. As per NCI-CTCAE version 4.03, Grade 1: loss of appetite without alteration in eating habits.
Time Frame: as for outcome 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Yes: Day 28: number analyzed (Participants) | 6
  Yes: Day 28 | 90.998 (72.5190)
  No: Day 28: number analyzed (Participants) | 28
  No: Day 28 | 81.971 (63.5134)
  Yes: Day 56: number analyzed (Participants) | 11
  Yes: Day 56 | 111.482 (54.9565)
  No: Day 56: number analyzed (Participants) | 30
  No: Day 56 | 76.606 (39.8971)
  Yes: Day 84: number analyzed (Participants) | 9
  Yes: Day 84 | 91.867 (57.5206)
  No: Day 84: number analyzed (Participants) | 35
  No: Day 84 | 76.520 (36.7957)

18. Secondary Outcome: Summary and Analysis of Trough Bosutinib Plasma Levels by Presence/Absence Grade 1: Vomiting
Description: Trough bosutinib plasma concentration is reported classified on basis of presence/ or absence of grade 1 vomiting as "Yes" and "No" at specified time points. As per NCI-CTCAE version 4.03, Grade 1: 1 - 2 episodes (separated by 5 minutes) in 24 hours.
Time Frame: as for outcome 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Yes: Day 28: number analyzed (Participants) | 7
  Yes: Day 28 | 58.826 (29.1613)
  No: Day 28: number analyzed (Participants) | 27
  No: Day 28 | 89.977 (69.3702)
  Yes: Day 56: number analyzed (Participants) | 11
  Yes: Day 56 | 87.135 (53.5627)
  No: Day 56: number analyzed (Participants) | 30
  No: Day 56 | 85.533 (44.5062)
  Yes: Day 84: number analyzed (Participants) | 10
  Yes: Day 84 | 90.030 (32.1444)
  No: Day 84: number analyzed (Participants) | 34
  No: Day 84 | 76.609 (43.8653)

19. Secondary Outcome: Summary and Analysis of Trough Bosutinib Plasma Levels by Presence/Absence Grade 1: Thrombocytopenia
Description: Trough bosutinib plasma concentration is reported classified on basis of presence/ or absence of grade 1 thrombocytopenia as "Yes" and "No" at specified time points. As per NCI-CTCAE version 4.03, Grade 1: platelet count decreased: 75.0 - 50.0*10^9/L.
Time Frame: as for outcome 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
ng/mL
  Yes: Day 28: number analyzed (Participants) | 3
  Yes: Day 28 | 80.167 (46.6352)
  No: Day 28: number analyzed (Participants) | 31
  No: Day 28 | 83.893 (66.1379)
  Yes: Day 56: number analyzed (Participants) | 5
  Yes: Day 56 | 87.700 (35.9669)
  No: Day 56: number analyzed (Participants) | 36
  No: Day 56 | 85.722 (48.0957)
  Yes: Day 84: number analyzed (Participants) | 3
  Yes: Day 84 | 75.067 (33.1815)
  No: Day 84: number analyzed (Participants) | 41
  No: Day 84 | 79.995 (42.4024)

20. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs): National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) (Version 4.03) Grade 3 or Higher
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. The severity was graded by NCI CTCAE v.4.03. Grade 1 was mild AE. Grade 2 was moderate AE. Grade 3 was severe AE. Grade 4 was life-threatening consequences and urgent intervention indicated AE. Grade 5 was death related to AE. Number of participants with Grade 3 or higher AEs are reported.
Time Frame: From first dose and up to 28 days after the last dose of study drug (maximum up to 45 months)
Population: As-treated population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Participants | 49

21. Secondary Outcome: Number of Participants With Laboratory Abnormalities, Chemistry: National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) (Version 4.03) Grade 3 or 4
Description: Laboratory parameters include: Alanine aminotransferase (ALT) increased: Grade 3: >5.0-20.0*upper limit of normal (ULN),Grade 4:>20.0*ULN, Alkaline phosphatase (ALP) increased: Grade 3: >5.0 - 20.0 x ULN, Grade 4: >20.0 x ULN, Aspartate aminotransferase (AST) increased: Grade 3: >5.0 - 20.0 *ULN, Grade 4: >20.0*ULN. Blood bilirubin increased:Grade 3:>3.0 - 10.0*ULN,Grade 4: >10.0*ULN, creatine phosphokinase (CPK) increased: Grade 3: >5*ULN-10*ULN, Grade 4: >10*ULN, Hyperglycemia: Grade 3: >250-500 milligrams/deciliter (mg/dL), Grade 4: >500 mg/dL. Hypermagnesemia: Grade 3: >3.0-8.0 mg/dL, Grade 4: >8.0 mg/dL, Hypokalemia: Grade 3: <3.0-2.5 millimoles/ liter (mmol/L), Grade 4:<2.5 mmol/L); Hyponatremia: Grade 3: <130-120 mmol/L, Grade 4: <120 mmol/L. Hypophosphatemia: Grade 3: <2.0-1.0 mg/dL, Grade 4: <1.0 mg/dL. Lipase increased: Grade 3:>2.0-5.0*ULN, Grade 4: >5.0*ULN. Serum amylase increased: Grade 3: >2.0 - 5.0*ULN, Grade 4: >5.0* ULN.
Time Frame: From first dose and up to 28 days after the last dose of study drug (maximum up to 45 months)
Population: As-treated population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Participants
  ALT increased | 30
  ALP increased | 1
  AST increased | 16
  Blood bilirubin increased | 1
  CPK increased | 3
  Hyperglycemia | 2
  Hypermagnesemia | 1
  Hypokalemia | 2
  Hyponatremia | 3
  Hypophosphatemia | 3
  Lipase increased | 14
  Serum amylase increased | 1
  Creatinine increased | 0
  Hypercalcemia: number analyzed (Participants) | 59
  Hypercalcemia | 0
  Hyperkalemia | 0
  Hypernatremia | 0
  Hypoalbuminemia | 0
  Hypocalcemia: number analyzed (Participants) | 59
  Hypocalcemia | 0
  Hypoglycemia | 0
  Hypomagnesemia | 0

22. Secondary Outcome: Number of Participants With Laboratory Abnormalities, Hematology: National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) (Version 4.03) Grade 3 or 4
Description: Laboratory parameters include: Anemia: Grade 3: hemoglobin (Hgb) <8.0 g/dL, Grade 4: Life-threatening consequences; urgent intervention indicated, Lymphocyte count decreased: Grade 3: <500 - 200/millimeter(mm)^3, Grade 4: <200/mm^3, Neutrophil count decreased: Grade 3: <1000 - 500/mm^3, Grade 4: <500/mm^3, Platelet count decreased: Grade 3: <50.0 - 25.0*10^9 /L, Grade 4: <25.0*10^9 /L. White blood cell decreased: Grade 3: <2.0 - 1.0*10^9 /L, Grade 4: <1.0*10^9 /L. Only those rows in which at least 1 participant had data were reported.
Time Frame: From first dose and up to 28 days after the last dose of study drug (maximum up to 45 months)
Population: As-treated population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Participants
  Anemia | 4
  Lymphocyte count decreased | 14
  Neutrophil count decreased | 9
  Platelet count decreased | 6
  White blood cell decreased | 2

23. Secondary Outcome: Number of Participants With Laboratory Abnormalities, Coagulation: National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) (Version 4.03) Grade 3
Description: Coagulation parameters include: APTT prolonged (Grade 3: >2.5*ULN and hemorrhage), and INR increased (Grade 3 >2.5*ULN).
Time Frame: From first dose and up to 12 March 2019; maximum of 22 months, approximately
Population: As-treated population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Participants
  Activated partial thromboplastin time | 0
  INR increased: number analyzed (Participants) | 56
  INR increased | 0

24. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Findings
Description: Vital signs included: body weight Increase >= 10% change from baseline and Decrease >= 10% change from baseline, systolic blood pressure in millimeters of mercury (mmHg): <80 mmHg and >210 mmHg, diastolic blood pressure in mmHg: <40 mmHg and >130 mmHg, heart rate in beats per minute (bpm): <40 bpm and >150 bpm, temperature in degree Celsius (C): <32 and >40 degree C.
Time Frame: From first dose and up to 28 days after the last dose of study drug (maximum up to 45 months)
Population: As-treated population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Participants
  Body weight: Increase >= 10% change from baseline: number analyzed (Participants) | 58
  Body weight: Increase >= 10% change from baseline | 12
  Body weight: Decrease >= 10% change from baseline: number analyzed (Participants) | 58
  Body weight: Decrease >= 10% change from baseline | 2
  Systolic blood pressure: <80 mmHg: number analyzed (Participants) | 58
  Systolic blood pressure: <80 mmHg | 0
  Systolic blood pressure: >210 mmHg: number analyzed (Participants) | 58
  Systolic blood pressure: >210 mmHg | 0
  Diastolic blood pressure: <40 mmHg: number analyzed (Participants) | 58
  Diastolic blood pressure: <40 mmHg | 1
  Diastolic blood pressure: >130 mmHg: number analyzed (Participants) | 58
  Diastolic blood pressure: >130 mmHg | 0
  Heart rate: <40 bpm: number analyzed (Participants) | 58
  Heart rate: <40 bpm | 0
  Heart rate: >150 bpm: number analyzed (Participants) | 58
  Heart rate: >150 bpm | 0
  Temperature: <32 C | 0
  Temperature: >40 C | 1

25. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: ECG parameters included: QTc corrected by Bazett's (QTcB) interval: >500 msec (milliseconds), QTc corrected by Fridericia's (QTcF) interval: >500 msec and >450 msec (men) or >470 msec (women).
Time Frame: From first dose and up to 28 days after the last dose of study drug (maximum up to 45 months)
Population: As-treated population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Participants
  QTcB interval: >500 msec | 0
  QTcF interval: >500 msec | 0
  QTcF interval: >450 msec (Men) or >470 msec (Women) | 1

26. Secondary Outcome: Number of Participants Assessed for Left Ventricular Ejection Fraction
Description: Interpretation categories included: a) normal, b) abnormal, not clinically significant and c) abnormal, clinically significant.
Time Frame: At end of treatment for patients who discontinued treatment post initial dose (up to 12 March 2019)
Population: As-treated population included all enrolled participants who received at least 1 dose of study treatment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 18
Participants
  Normal | 15
  Abnormal, not clinically significant | 3
  Abnormal, Clinically Significant | 0

27. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) at Months 3, 6, 9 and 18
Description: A MMR is defined as less than or equal to (<=) 0.1 percent (%) BCR-ABL transcripts on the international scale (IS), corresponding to a >=3-log reduction from standardized baseline with at least 3000 ABL assessed by the central laboratory. The MMR value counted only if the response was demonstrated at the designated visit; any MMR gained and lost, or never achieved at or before the designated visit was considered as non-responder.
Time Frame: Month 3, 6, 9 and 18
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants
  Month 3 | 10.0 [3.6 to 16.4]
  Month 6 | 50.0 [39.4 to 60.6]
  Month 9 | 53.3 [42.7 to 63.9]
  Month 18 | 61.7 [51.3 to 72.0]

28. Secondary Outcome: Percentage of Participants With Molecular Response 1 (MR1) at Month 3
Description: MR1 is defined as <= 10% BCR-ABL with a minimum of 3,000 ABL transcripts assessed by the central laboratory.
Time Frame: Month 3
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 80.0 [71.5 to 88.5]

29. Secondary Outcome: Percentage of Participants With Molecular Response 2 (MR2) at Month 6
Description: MR2 is defined as <= 1% BCR-ABL with a minimum of 3,000 ABL transcripts assessed by the central laboratory.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 66.7 [56.7 to 76.7]

30. Secondary Outcome: Percentage of Participants With Molecular Response 4.0 (MR4.0) and Molecular Response 4.5 (MR4.5) at Months 3, 6, 9 and 12
Description: MR4.0 defined as either: detectable disease with <= 0.01% BCR-ABL with a minimum of 9,800 ABL transcripts assessed by the central laboratory, or undetectable disease in cDNA with a minimum of 9,800 ABL transcripts assessed by the central laboratory. MR4.5 defined as either: detectable disease with <= 0.0032% BCR-ABL with a minimum of 30,990 ABL transcripts assessed by the central laboratory or undetectable disease in cDNA with a minimum of 30,990 ABL transcripts assessed by the central laboratory. The MMR value counted only if the response was demonstrated at the designated visit; any MMR gained and lost, or never achieved at or before the designated visit was considered as non-responder.
Time Frame: Months 3, 6, 9 and 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants
  MR4.0: Month 3 | 0 [0.0 to 0.0]
  MR4.0: Month 6 | 18.3 [10.1 to 26.5]
  MR4.0: Month 9 | 25.0 [15.8 to 34.2]
  MR4.0: Month 12 | 31.7 [21.8 to 41.5]
  MR4.5: Month 3 | 0 [0.0 to 0.0]
  MR4.5: Month 6 | 8.3 [2.5 to 14.2]
  MR4.5: Month 9 | 16.7 [8.8 to 24.6]
  MR4.5: Month 12 | 21.7 [12.9 to 30.4]

31. Secondary Outcome: Cumulative Incidence of Major Molecular Response (MMR) at Month 36
Description: Percentage of participants with MMR at Month 36. Cumulative incidence of MMR was measured from first dose to the first date of response. Documented participants who did not have an MMR response were censored at the last molecular assessment. A MMR is defined as <=0.1% BCR-ABL transcripts on the international scale, corresponding to a >=3-log reduction from standardized baseline with at least 3000 ABL assessed by the central laboratory. Cumulative incidence: % of participants with event at month 36 adjusted for competing risk of treatment discontinuation without the event.
Time Frame: At Month 36
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 70.0 [60.3 to 79.7]

32. Secondary Outcome: Cumulative Incidence of Molecular Response 4.0 (MR4.0) at Month 36
Description: Percentage of participants with MR4.0 at month 36. Cumulative incidence of MR4.0, was measured from first dose to the first date of MR 4.0. Documented participants who did not have an MR4.0 response were censored at the last molecular assessment. MR4.0 defined as either 1) detectable disease with <=0.01% BCR-ABL IS or 2) undetectable disease in cDNA with a minimum number of 9800 ABL transcripts specified by the central laboratory. Cumulative incidence: % of participants with event at month 36 adjusted for competing risk of treatment discontinuation without the event.
Time Frame: At Month 36
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 50.0 [39.4 to 60.6]

33. Secondary Outcome: Cumulative Incidence of Molecular Response 4.5 (MR4.5) at Month 36
Description: Percentage of participants with MR4.5 at Month 36. Cumulative incidence of MR 4.5 was measured from first dose to the first date of MR 4.5. Documented participants who did not have an MR4.5 response were censored at the last molecular assessment. MR 4.5 defined as either 1) detectable disease with <=0.0032% BCR-ABL IS or 2) undetectable disease in cDNA with a minimum number of 30990 ABL transcripts specified by the central laboratory in the same volume of cDNA used to test for BCR-ABL. Cumulative incidence: % of participants with event at month 36 adjusted for competing risk of treatment discontinuation without the event.
Time Frame: At Month 36
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 46.7 [36.1 to 57.3]

34. Secondary Outcome: Cumulative Incidence of Complete Cytogenetic Response (CCyR) at Month 36
Description: Percentage of participants with CCyR at Month 36. Cumulative incidence of CCyR, was measured from first dose to the first date of CCyR. Documented participants who did not have a CCyR response were censored at the last cytogenetic assessment. CCyR was defined as absence of detectable Philadelphia chromosome positive cells. CCyR was achieved when there were "0" Philadelphia chromosome positive metaphases among at least 20 metaphases from a bone marrow sample or when MMR was achieved if no bone marrow analysis was performed. Cumulative incidence: % of participants with event at month 36 adjusted for competing risk of treatment discontinuation without the event.
Time Frame: At Month 36
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 80.0 [69.8 to 87.1]

35. Secondary Outcome: Percentage of Participants With Cumulative Complete Haematological Response (CHR)
Description: CHR is based on peripheral blood assessment: WBC <=10*10^9/L, basophils <5% in blood, no myelocytes, promyelocytes, myeloblasts in the blood differential, platelet count <450* 10^9/L, spleen non-palpable. In the absence of extramedullary disease info, it was assumed that spleen was non-palpable. If CHR could not be assessed due to one or more missing components of CHR and participant had a MMR or a CCyR and all assessed components of CHR were within appropriate limits, then CHR was imputed using CCyR or MMR. CHR must be of at least 4 weeks in duration and confirmed by 2 assessments at least 4 weeks apart.
Time Frame: Up to Month 36
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | 91.7 [85.8 to 97.5]

36. Secondary Outcome: Cumulative Incidence of Transformation to Accelerated Phase (AP) and Blast Phase (BP) at Month 36
Description: Percentage of participants with transformation to AP and BP at Month 36. Transformation to AP or to BP CML defined as the time from first dose to the first date of transformation to accelerated phase or to blast phase CML. Documented participants who did not progress to AP or BP were censored at the last hematologic assessment. The transformation to AP or to BP was counted while participants were on treatment up to 28 days after last dose. Cumulative incidence: % of participants with event at month 36 adjusted for competing risk of treatment discontinuation without the event.
Time Frame: At Month 36
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 60
Percentage of participants | NA [NA to NA] — Number and 90% CI was not estimable as there were no participants with events.

37. Secondary Outcome: Number of Participants With BCR-ABL Mutation at Treatment Discontinuation
Description: Mutation analysis was performed in case of either lack of response, suboptimal response or loss of response, or at the End of Treatment/Withdrawal visit.
Time Frame: Maximum up to 44 months of treatment
Population: The modified as-treated population included all enrolled participants with Philadelphia chromosome positive CP CML harboring b2a2 and/or b3a2 transcripts who received at least 1 dose of study treatment. Here, ''Overall Number of Participants Analyzed'' signifies participants with mutation testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 24
Participants | 0

ADVERSE EVENTS:
Time Frame: From first dose and up to 28 days after the last dose of study drug (maximum up to 45 months)
Description: The total number of deaths occurring during study, from first dose and up to end of the study are reported for all treated participants and includes deaths which occurred after 28 days post last study drug dose. Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety population evaluated.
Arm/Group | Bosutinib
All-Cause Mortality (participants affected / at risk) | 2/60
Serious Adverse Events (participants affected / at risk) | 14/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=60)
Diabetic retinopathy (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 2
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Influenza (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=60)
Anaemia (Blood and lymphatic system disorders) | 10
Lymphopenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 52
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 16
Pyrexia (General disorders) | 15
Liver disorder (Hepatobiliary disorders) | 7
Influenza (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 23
Upper respiratory tract infection (Infections and infestations) | 8
Alanine aminotransferase increased (Investigations) | 33
Amylase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 28
Blood alkaline phosphatase increased (Investigations) | 16
Blood creatine phosphokinase increased (Investigations) | 6
Gamma-glutamyltransferase increased (Investigations) | 11
Lipase increased (Investigations) | 17
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 13
White blood cell count decreased (Investigations) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 4
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 18
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Stomatitis (Gastrointestinal disorders) | 6
Gastroenteritis (Infections and infestations) | 5
Blood creatinine increased (Investigations) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT03128411/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT03128411/SAP_001.pdf